CLINICAL TRIAL: NCT02531529
Title: Dexmedetomedine Infusion Versus Fentanyl Infusion for Donor Anlgesia During Living Donor Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LTx 1
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Donor Hepatectomy
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- D group (Experimental): intraoperative dexmedetomedine infusion
  Interventions: Drug: dexmedetomedine
- F group (Sham Comparator): Intraoperative fentanyl infusion
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: dexmedetomedine — intraoperative infusion
  Arms: D group
Drug: Fentanyl
  Arms: F group

SUMMARY:
To compare between the analgesic effect of dexmedetomedine infusion versus Fentanyl infusion during donor hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* donors of living donor liver transplantation

Exclusion Criteria:

* patient refusal Known allergy to dexmedetomedine

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
postoperative VAS scale | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dkahleya, Egypt